CLINICAL TRIAL: NCT05061108
Title: Linkage, Empowerment, and Access to Prevent Hypertension (LEAP-HTN)
Brief Title: Linkage, Empowerment, and Access to Prevent Hypertension
Acronym: LEAPHTN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Phillip Levy, Professor, Assistant Vice President for Translational Sciences and Clinical Research Innovation, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 878605
Record Dates: First submitted 2021-09-07; First posted 2021-09-29 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Blood Pressure; Cardiovascular Disease Other
Keywords: Health Disparities; African American; Prevention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Randomized selection of recruited participants that will receive intervention
  Interventions: Behavioral: PAL2
- Control (No Intervention): Randomized selection of recruited participants that will not receive intervention

INTERVENTIONS:
Behavioral: PAL2 — Community health worked based intervention to mitigate psychosocial and life circumstance barriers to optimize health promotion coupled with high blood pressure and lifestyle disease state education
  Other Names: Pragmatic personalized, adaptable approach to lifestyle and life circumstance
  Arms: Intervention

SUMMARY:
Brief Summary:

Black adults have a higher incidence of hypertension (HTN) and a greater risk of HTN-related cardiovascular disease (CVD) compared with White adults. Even mild elevations in blood (BP) above 115/75 mm Hg are associated with increased CVD risk. Accordingly, emphasis is being placed on early interventions for high BP, particularly in those who are low cardiovascular risk(systolic BP 110-139 and diastolic BP < 90 mm Hg), for participants lifestyle modification is recommended. Although lifestyle modifications are effective to lower BP, implementation is suboptimal in Black communities, especially those participants residing in low-income urban settings. Pervasive negative social determinants of health (SDoH), such as poor access to healthcare, food insecurity, limited availability of healthy foods, lack of safe places to engage in physical activity, and low health literacy are major drivers of inequities in HTN and a critical barrier to implementation of recommended lifestyle modifications in Black communities. To achieve health equity, effective strategies must address negative SDoH that are root causes of racial disparities in health outcomes as clearly demonstrated by the coronavirus disease (COVID-19) pandemic. Predominantly Black cities like Detroit, Michigan, where the mortality rate from heart disease is nearly twice the national average, have been devastated by COVID-19. To address this, the investigators developed an innovative mobile health unit (MHU) program that uses geospatial health and social vulnerability data to direct deployment of testing and vaccination services to communities with highest needs. Since April 2020, the investigators conducted 500 events with 220 community partners where 40,000 people have been tested or vaccinated for COVID in MHUs.

Using a hybrid type I effectiveness-implementation design in the proposed Linkage, Empowerment, and Access to Prevent Hypertension (LEAP-HTN) study, the investigators will implement a novel approach that links low cardiovascular risk Black adult participants without stage-2 hypertension to collaborative care delivered in deprived neighborhoods by community health workers (CHWs) using a personalized, adaptable approach to lifestyle and life circumstance (PAL2) intervention. The investigators will leverage our MHU program, layering on top of existing services to streamline access for screening, recruitment and all ongoing follow-up throughout the study period. Our specific aims are:

AIM 1: To compare the effect of PAL2 intervention versus usual care (MHU engagement without PAL2) on systolic BP reduction and prevention of stage 2 HTN (systolic BP ≥ 140 mm Hg and/or diastolic BP >90 mm Hg) among 500 Black adults with baseline untreated systolic BPs below stage 2 (ranging 110-139 mm Hg) and a diastolic BP < 90 mm Hg.

Hypothesis (H) 1a: Systolic BP (primary outcome) will be reduced more in those randomized to PAL2 intervention versus usual care at 6 and 12 months.

H1b: Diastolic BP levels and the incidence of stage 2 HTN (systolic BP ≥ 140 mm Hg and/or diastolic BP >90 mmm Hg) at 6 and 12 months (secondary outcomes) will be lower in participants randomized to the PAL2 intervention versus usual care.

AIM 2: To use the RE-AIM framework to assess the reach, adoption, effectiveness, sustainability and cost of LEAP-HTN at 12 months post-randomization.

H2a: The rates of adoption and sustainability of the PAL2 intervention will increase from baseline to 12 and up to 24 months in subjects with available data, respectively.

H2b: PAL2 intervention will be more cost-effective than usual care at 12 months and projected to be more cost-effective at 10 years.

Health Equity Impact: Targeted deployment of MHUs and PAL2 can mitigate several key adverse SDoH. LEAP-HTN contributes to the RESTORE Network by testing a sustainable and scalable approach to advance health equity and prevent HTN in Black adults participants. If successful, the use of MHU can be easily implemented in similar urban Black communities across the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identification as Black, age ≥18 years, living in the Detroit-area
2. Systolic BP 110-139 and diastolic BP <90 mm Hg upon screening
3. Not currently taking medications for HTN
4. Low cardiovascular risk as defined by 2017 AHA/ACC HTN guidelines (no diabetes, no chronic kidney disease, no established ASCVD
5. 10-year ASCVD risk <10% if systolic BP is in stage-1 hypertension range (130-139 mm Hg and < 65 years old

Exclusion Criteria:

1. Any clinical cardiovascular disease (e.g., coronary artery disease, heart failure, stroke, arrhythmia)
2. Chronic kidney disease or glomerular filtration rate <60 ml/min on screening laboratory testing
3. Diabetes or HbA1c ≥ 6.5% on screening laboratory testing
4. LDL-C ≥ 190 mg/dL on screening laboratory testing (on or off medications)
5. ASCVD risk score calculated ≥ 10% for 10 years by clinical calculator on screening (if stage-1 systolic HTN only)2
6. Inability or not willing to follow-up with PAL2 research or usual care limb and at 6 & 12-months at the MHU
7. Taking any medications for diabetes, heart disease or kidney disease. Cholesterol medication is not an exclusion
8. Inability to understand and sign informed consent

10. Chronic condition (e.g., cancer) with a potential life expectancy < 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Systolic BP levels will be significantly lower (by ≥4 mm Hg) in participants randomized to the PAL2 (active) intervention versus usual care (control) over the first 12 months of the trial | 12 months
  Resting seated systolic BP will be measured in the dominant upper arm by validated automated BP monitors using a standardized protocol in accordance with the methods in the 2017 American College of Cardiology (ACC)/American Heart Association (AHA) Hypertension guidelines. BP outcomes will be checked during months 6 and 12 of the trial

SECONDARY OUTCOMES:
PAL2 (active) intervention will lower diastolic BP compared to usual care (control). | 12 Months
  Resting seated diastolic BP will be measured in the dominant upper arm by validated automated BP monitors using a standardized protocol in accordance with the methods in the 2017 ACC/AHA Hypertension guidelines. BP outcomes will be checked during months 6 and 12 of the trial
PAL2 (active) intervention will lower the incidence of stage-1 hypertension compared to the control group over 1 year | 12 months
  Resting seated systolic and diastolic BPs will be measured in the dominant upper arm by validated automated BP monitors using a standardized protocol in accordance with the methods in the 2017 ACC/AHA Hypertension guidelines. BP outcomes will be checked during months 6 and 12 of the trial. Stage-1 hypertension is defined as a systolic BP ≥130 mm Hg and/or a diastolic BP ≥80 mm Hg.
The rates of adoption and sustainability of the PAL2 intervention will increase from baseline to 12 and 24 months, respectively. | 24 months
  Standardized surveys regarding the rate of compliance with the PAL2 intervention will be delivered at 6,12 and 24 months of the trial. These rates will be higher at 12 and 24 months versus 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne Health Mobile Units, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided